CLINICAL TRIAL: NCT05639387
Title: TMS as a Tool for the Evaluation of Neuromodulatory Effects of Transcutaneous Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/0988
Record Dates: First submitted 2022-11-09; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Each participant will complete 2 sessions at least one week apart, one with active tVNS and one with sham tVNS.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group of healthy volunteers (part I) (Experimental): Participants will undergo active tVNS.
  Interventions: Procedure: actual tVNS
- Group of healthy volunteers (part II) (Sham Comparator): Participants will undergo sham tVNS.
  Interventions: Procedure: sham tVNS

INTERVENTIONS:
Procedure: actual tVNS — Active tVNS (stimulation on cymba conchae --> nervus vagus stimulation)
  Arms: Group of healthy volunteers (part I)
Procedure: sham tVNS — Sham tVNS (stimulation on earlobe --> no nervus vagus stimulation)
  Arms: Group of healthy volunteers (part II)

SUMMARY:
Transcutaneous vagus nerve stimulation (tVNS) has been investigated as a potential treatment for epilepsy with inconsistent results. The combination of transcranial magnetic stimulation with electromyography (TMS-EMG) and electroencephalography (TMS-EEG) allows to investigate the neuromodulatory effect of interventions such as tVNS by evaluating changes in motor evoked potentials (MEPs) and TMS-evoked potentials (TEPs). The goal of this study is to objectively evaluate the effect of tVNS on cortical excitability with TMS-EMG and TMS-EEG. These findings are expected to provide insight in the mechanism of action and help identify more optimal stimulation paradigms.

In this prospective single-blind cross-over study, 15 healthy subjects will undergo active and sham tVNS during 60 minutes, using a maximum tolerated stimulation current. Single and paired pulse TMS will be delivered over the right-sided motor hotspot to evaluate MEPs and TEPs before and after the intervention.

DETAILED DESCRIPTION:
In the past two decades, vagus nerve stimulation (VNS)has become a valuable treatment option for patients with refractory epilepsy. However, VNS requires a surgical procedure associated with potential side effects. Therefore, the development of non-invasive devices that selectively target the vagus nerve fibers with a low risk profile has gained interest. Transcutaneous auricular VNS (tVNS) is such a non-invasive neurostimulation modality that targets the cutaneous receptive field of the auricular branch of the vagus nerve located in the outer ear. Up to date, tVNS has been investigated as a potential treatment for epilepsy with inconsistent results. The goal of this study is to investigate the effect of tVNS on cortical excitability. This will provide important insight into the underlying effects of this technique on brain neurophysiology. Cortical excitability will be investigated by combining transcranial magnetic stimulation with electromyography (TMS-EMG) and electroencephalography (TMS-EEG), evaluating changes in motor evoked potentials (MEPs) and TMS-evoked potentials (TEPs).

In this prospective, single-blind, cross-over study, we will include 15 healthy male participants. They will undergo a TMS safety screening (TSS) questionnaire and clinical neurological examination before inclusion. Each participant will complete 2 sessions at least one week apart, one with active tVNS and one with sham tVNS.

The intervention is tVNS by means of the Nemos® device which stimulates the cymba conchae at the outer ear. Stimulation parameters are set to a frequency of 25 Hz, a pulsewidth of 250 µs, 7 s ON, 18 s OFF. The output current is ramped up until the user feels a tingling sensation at the stimulation site, but should remain subthreshold to painful stimulation. Stimulation is delivered during 60 min.Sham stimulation is achieved by placing the electrode on the earlobe instead of the cymba conchae.

Before and after the intervention 120 single TMS pulses, 120 paired pulses with an interstimulus interval of 3ms and 120 paired pulses with an interstimulus interval of 100ms will be delivered over the right motor hotspot. MEPs will be measured at the left first dorsal interosseus muscle. TEPs will be measured using a 64-channel TMS-compatible electrode cap. MEPS and TEPS will be preprocessed offline in Matlab. TEP and MEP morphology ( amplitude and latency) will be evaluated before and after the intervention to investigate changes in cortical excitability.

ELIGIBILITY:
Inclusion Criteria:

* estimated IQ > 70
* healthy volunteer, taken from anamensis, clinical neurological examination and clinical estimation of researcher
* no history of central neurological condition
* no treatment with neurotropic drugs
* TMS safety screening questionnaire
* ICF signed

Exclusion Criteria:

* intracranial metal objects/materials (excl teeth fillings): vascular clips, shrapnell electrodes below stimulation area
* pacemaker, implanted defibrillator, permanent medication pump, cochlear implant or deep brain stimulation (DBS)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Measuring the electric activity of the brain evaluating changes in motor evoked potentials (MEPs) and TMS-evoked potentials (TEPs) during transcutaneous nervus vagus stimulation. | 60 minutes
  Using transcranial magnetic stimulation (TMS), the influence of the tVNS is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium